CLINICAL TRIAL: NCT06706804
Title: The Effect of Wiping Bath Training on Early Bathing, Body Temperature and Umbilical Cord Fall Time in Newborns: a Randomized Controlled Trial
Brief Title: The Effect of Wiping Bath Training on Early Bathing, Body Temperature and Umbilical Cord Fall Time in Newborns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çağla KILIÇ (Other)
Responsible Party: Sponsor-Investigator, Çağla KILIÇ, Research Assistant, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSÜ MIDWIFERY DEPARTMENT
Record Dates: First submitted 2024-11-15; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Wiping Bath; Education; Newborn
Keywords: Education; Newborn; Newborn bathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: (No Intervention): Pregnant women in the control group will be subjected to the routine hospital protocol and will not be subjected to any other intervention. In the pregnancy schools of the hospitals, they are verbally told not to wash and wipe their babies before the umbilical cord falls off. After the training, pregnant women will be given a home follow-up form to record the first bath time of their babies after birth, the umbilical cord fall time and the body temperature of their babies (before bathing, immediately after bathing and 10 minutes after bathing) and will be told how to fill it out.
- Wipe Bathing (Experimental): In groups of 2-3 pregnant women in this group, the researcher will explain the stages of newborn wiping bath application on the newborn model, and then the pregnant women will individually apply the bath on the model. The trainings will be held in the pregnant school at the appropriate hours, or in an empty room determined by the hospital administration if there is another planned training in the pregnant school. In the wiping bath training, for genital area cleaning based on the gender of newborns, women will be provided to perform the procedure on the model appropriate to the gender of their babies. After the training, pregnant women will be given a home follow-up form to record the first bath time of their babies after birth, the umbilical cord fall time and the body temperature of their babies (before bathing, immediately after bathing and 10 minutes after bathing) and will be told how to fill it out.
  Interventions: Behavioral: Wipe Bathing

INTERVENTIONS:
Behavioral: Wipe Bathing — In groups of 2-3 pregnant women in this group, the researcher will explain the stages of newborn wiping bath application on the newborn model, and then the pregnant women will individually apply the bath on the model. The trainings will be held in the pregnant school at the appropriate times, or in an empty room determined by the hospital administration if there is another planned training in the pregnant school. In the wiping bath training, women will be provided to perform the procedure on the model appropriate to the gender of their babies for genital area cleaning based on the gender of newborns. After the training, pregnant women will be given a home follow-up form to record the first bath time of their babies after birth, the umbilical cord fall time and the body temperature of their babies (before bathing, immediately after bathing and 10 minutes after bathing) and will be told how to fill it out.
  Arms: Wipe Bathing

SUMMARY:
The aim of this study is to examine the effects of wiping bath training on early bathing, body temperature and umbilical cord shedding time in newborns. This study was planned in a randomized controlled experimental research design. The study will be conducted with pregnant women who applied to the pregnancy schools of Kahramanmaraş Necip Fazıl City Hospital Gynecology and Obstetrics Additional Service building. When calculating the sample size, a similar study previously conducted on the subject was taken as a reference and the G*Power 3.1.9.7 program was used (Ayyıldız et al, 2015). In the calculation made; the sample size of the study was found to be at least 36, and considering the parametric distribution, it was planned to complete the study with a total of 60 people, 30 in each group. Considering the possible case losses (10%), it is planned to include a total of 66 women (intervention group: 33, control group: 33). In the study, women will be assigned to groups according to the previously determined randomization number sequences, and then the Pregnant Information Form will be filled out by the participants using the face-to-face interview method. The determined practices will be carried out according to the group to which the participants are assigned. The hospital's pregnancy information class will be used for the training, and if there is another planned training in the pregnancy school, an empty room determined by the hospital administration will be used. The pregnant women in the intervention group will be explained the newborn wiping and bathing application stages by the researcher in groups of 2-3 people on a newborn model, and then the pregnant women will be asked to apply the bath individually on the model. The pregnant women in the control group will be subject to routine hospital protocol and no other intervention will be made. After the birth, the participants will be called by phone and the "Newborn Characteristics Information Form" will be filled out by phone and the participants will be asked to provide information by phone message after the umbilical cord falls off. After the umbilical cord falls off, the participants will be called by phone and the first bath time, umbilical cord falling off time and the body temperature of their babies (before the bath, immediately after the bath and 10 minutes after the bath) will be recorded by asking the mothers on the given follow-up form.

DETAILED DESCRIPTION:
This study will be conducted in a randomized controlled experimental research design.

ELIGIBILITY:
Inclusion Criteria

* Infants of women who can speak and understand Turkish,
* who are literate, who are between 38-40 weeks of gestation,
* who have a healthy pregnancy,
* who can be followed up in the postpartum period by obtaining contact information, -who have a thermometer that can measure their baby's temperature at home, ---
* whose mothers do not have chronic-systemic diseases, hepatitis, acquired immunodeficiency syndrome and genital infections,
* who voluntarily agree to participate in the study and give written informed consent will be included in the study.

Exclusion Criteria

* Newborns with a gestational age below 37 weeks,
* birth weight below 2500 grams,
* premature rupture of membranes in the mother,
* congenital defects,
* need for intensive care or hospitalization,
* impaired skin integrity or skin problems and newborns whose mothers could not be contacted after birth will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Early Bathing Rate | 2 weeks after birth
  Early Bathing Rate will be determined using the Newborn Home Monitoring Form. This form was developed by the researchers to ensure that mothers record information about the newborn regularly at home and to collect the necessary data for the study. The form will be given to the mothers after the bathing training and they will be asked to fill it in at home. Mothers will be asked to record the baby's first bath time on this form. Baths before 24 hours postpartum will be considered early bathing.
Newborn Body Temperature | 2 weeks after birth
  The body temperature of the newborn will be determined using the Newborn Home Monitoring Form. This form was developed by the researchers to ensure that mothers record information about the newborn regularly at home and to collect the necessary data for the study. The form will be given to the mothers after the bathing training and they will be asked to fill it in at home. Mothers will be asked to record their body temperature measurements before, immediately after and 10 minutes after the baby's first bath on this form. Body temperature will be calculated as mean±SD.
The duration of umbilical cord fall | 2 weeks after birth
  The duration of umbilical cord fall will be determined using the Newborn Home Monitoring Form. This form was developed by the researchers to ensure that mothers record information about the newborn regularly at home and to collect the necessary data for the study. The form will be given to the mothers after the bathing training and they will be asked to fill it in at home. Mothers will be asked to write the date of the umbilical cord drop on this form. Duration of umbilical cord fall will be calculated as mean±SD.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta P, Nagesh K, Garg P, Thomas J, Suryawanshi P, Sethuraman G, Hazarika RD, Verma RJ, Kumar CS, Kumari S, Taneja S, Chavhan V, Thakor P, Pandita A. Evidence-Based Consensus Recommendations for Skin Care in Healthy, Full-Term Neonates in India. Pediatric Health Med Ther. 2023 Aug 25;14:249-265. doi: 10.2147/PHMT.S414091. eCollection 2023. PMID 37654800
- [Background] Gozen D, Caka SY, Besirik SA, Perk Y. First bathing time of newborn infants after birth: A comparative analysis. J Spec Pediatr Nurs. 2019 Apr;24(2):e12239. doi: 10.1111/jspn.12239. Epub 2019 Mar 19. PMID 30887671